Official Title: A Phase 1, Open-label, Positron Emission Tomography Study in Healthy Subjects to Determine the Relationship Between Plasma Concentration and Target Occupancy of ASN51 Following Repeated Oral Doses

NCT ID: NCT05725005

**Document Date:** SAP Version 1.1: 13 June 2023

## **Statistical Analysis Plan**

Clinical trial protocol title: A phase 1, open-label, positron emission tomography

study in healthy subjects to determine the relationship between plasma concentration and target occupancy of

ASN51 following repeated oral doses.

HMR code: 22-012

Sponsor code: ASN51-103

IRAS number: 1006677

CRO details: HMR

Cumberland Avenue London NW10 7EW

Sponsor details: Asceneuron S.A.

EPFL Innovation Park, Bâtiment B 1015 Lausanne, Switzerland, CH-1015

Issued: 13 June 2023

Version: 1.1

Based on: Protocol version 2, dated 23 January 2023

Prepared by:

# **Version control history**

| Version | Reason for change |
|---|---|
| 1, dated 22 May 2023 | N/A |
| 1.1, dated 12 Jun 2023 | Updated a formatting error in section 12.1 in relation to |
| | Appendix A and Appendix B. Removed column "Study |
| | Day" from T14.2.1.1 as not required. |

# **Table of Contents**

| VER | SION ( | CONTROL HISTORY | 1 |
|-----|--------|-------------------------------------------------------|----|
| 1 | LIST | OF ABBREVIATIONS | 5 |
| 2 | SIGN | NATURES | 7 |
| 3 | INTE | RODUCTION | 8 |
| 4 | STU | DY OBJECTIVE(S) AND ENDPOINT(S) | 8 |
| | 4.1 | Study objective(s) | 8 |
| | | 4.1.1 Primary objective(s) | 8 |
| | | 4.1.2 Secondary objective(s) | 8 |
| | 4.2 | Study endpoint(s) | 9 |
| | | 4.2.1 Primary endpoint(s) | 9 |
| | | 4.2.2 Secondary endpoint(s) | 9 |
| | 4.3 | Statistical hypotheses | 9 |
| 5 | STU | DY DESIGN | 10 |
| | | 5.1.1 PBMC-only subjects | 10 |
| | | 5.1.2 PET subjects | 10 |
| 6 | TIM | E AND EVENTS TABLE | 11 |
| 7 | PLA: | NNED ANALYSES | 11 |
| | 7.1 | Interim analyses | 12 |
| | 7.2 | Final analysis | 12 |
| | | 7.2.1 Persons responsible for analysis | 12 |
| 8 | SAM | IPLE SIZE CONSIDERATIONS | 12 |
| | 8.1 | Sample size assumptions | 12 |
| 9 | ANA | LYSIS POPULATIONS | 12 |
| | 9.1 | Analysis datasets | 13 |
| 10 | TRE | ATMENT COMPARISONS | 13 |
| 11 | GEN | ERAL CONSIDERATIONS FOR DATA ANALYSES | 13 |
| | 11.1 | Data display treatment and other subgroup descriptors | 13 |
| | 11.2 | Conventions for summary statistics and data displays | |
| 12 | DAT | A HANDLING CONVENTIONS | |
| | 12.1 | Premature withdrawal and missing data | |
| | 12.2 | Derived and transformed data | |
| | 12.3 | Assessment windows | |
| | 12.4 | Vital signs reference ranges | |
| 13 | | DY POPULATION | |
| | ~ | | |

| | 13.1 | Disposition of subjects | 15 |
|---|---|---|---|
| | 13.2 | Protocol deviations | 15 |
| | 13.3 | Demographic and baseline characteristics | 16 |
| | 13.4 | Treatment compliance | 16 |
| 14 | SAFE | TY ANALYSES | 16 |
| | 14.1 | Extent of exposure | 16 |
| | 14.2 | Adverse events | 16 |
| | 14.3 | Deaths, serious adverse events and other significant adverse events | 17 |
| | 14.4 | Adverse events leading to withdrawal from the study | 17 |
| | 14.5 | Clinical laboratory evaluations | 17 |
| | 14.6 | Other safety measures | 17 |
| | | 14.6.1 Vital signs | 17 |
| | | 14.6.2 ECG | 17 |
| | | 14.6.3 Physical examination | |
| | | 14.6.4 Columbia-Suicide Severity Rating Scale (C-SSRS) | |
| 15 | PHAR | RMACOKINETIC ANALYSES | 18 |
| | 15.1 | Pharmacokinetic concentration data | 18 |
| | 15.2 | Pharmacokinetic parameters | 19 |
| 16 | PHAR | RMACODYNAMIC ANALYSES | 19 |
| 17 | CHAN<br>19 | NGES FROM THE PROTOCOL SPECIFIED STATISTICAL A | NALYSIS |
| 18 | REFE | RENCES | 20 |
| 19 | ATTA | CHMENTS | 20 |
| | 19.1 | Table of contents for data display specifications | 20 |
| | 19.2 | Data Display Specifications | 25 |
| | | 19.2.1 Table Outlines | 25 |
| | | 19.2.2 Figure Outlines | 38 |
| | | 19.2.3 Listing Outlines | 43 |
| APPE | ENDIX | A: LABORATORY TESTS WITH DIFFERENT RANGES | 51 |
| APPE | ENDIX | B: PHARMACOKINETIC ANALYSIS | 51 |
| 1 | CALC | CULATION METHODS | 51 |
| | 1.1 | Data Handling Conventions | 51 |
| | | 1.1.1 Actual v Planned Times | 51 |
| | | 1.1.2 Missing and BQL Concentrations | 51 |
| | 1.2 | AUC Calculations | 52 |

| A DI | PENDI | X C: SAMPLE PAGE LAYOUT | 56 |
|------|-------|-----------------------------|----|
| | 2.1 | Plasma Parameters | 54 |
| 2 | PAR | AMETER DEFINITIONS | 54 |
| | 1.5 | Achievement of Steady-State | 53 |
| | 1.4 | Observed v Predicted Values | 53 |

#### 1 List of abbreviations

 $\lambda_z$  Terminal rate constant

AE Adverse event

ANOVA Analyses of variance ANCOVA Analysis of covariance

AUC Area under concentration-time curve
AUC<sub>inf</sub> AUC from time zero to infinity
AUC for the dosing interval

AUC from time zero to last measurable concentration
%AUC<sub>extrap</sub>
%AUC<sub>extrap</sub>
AUC from time zero to last measurable concentration
Percentage of AUC<sub>inf</sub> extrapolated from from tlast to infinity

BMI Body mass index

BQL Below the limit of quantification

CI Confidence interval

CL<sub>ss</sub>/F Apparent total body clearance at steady state

C<sub>max</sub> Maximum plasma concentration

Ctrough Trough concentration
CRF Case report form
CSR Clinical study report

C-SSRS Columbia-Suicide Severity Rating Scale

CV Coefficient of variation CVb Between-subject CV ECG Electrocardiogram

FDA Food and Drug Administration

HR Heart rate

ICH International Conference on Harmonization

IV Intravenous

LSM Least Square Means

MedDRA Medical Dictionary for Regulatory Activities

N Number of subjects

n Number of observations used in analysis
PBMC Peripheral blood mononuclear cell
PET Positron emission tomography

PD Pharmacodynamic PK Pharmacokinetic(s)

PR Portion of the ECG from the beginning of the P wave to the beginning of

the QRS complex, representing atrioventricular node function.

QD Once a day

QRS The QRS complex of the ECG reflects the rapid depolarization of the right

and left ventricles

QT Portion of the ECG between the onset of the Q wave and the end of the T

wave, representing the total time for ventricular depolarization and

repolarization.

QTc Corrected portion of the ECG between the onset of the Q wave and the end

of the T wave, representing the total time for ventricular depolarization and

repolarization

OTcF OTc interval with Fridericia's correction method

 $\begin{array}{ll} R_{ac(AUC)} & Accumulation\ ratio\ for\ AUC \\ R_{ac(Cmax)} & Accumulation\ ratio\ for\ Cmax \end{array}$ 

RO Receptor Occupancy

| RR | Portion of the ECG between consecutive R waves, representing the ventricular rate |
|---|---|
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SRG | Safety Review Grouip |
| $\mathbf{t}_{1/2}$ | Terminal elimination half-life |
| TEAE | Treatment-emergent adverse event |
| $t_{max}$ | Time to maximum plasma concentration |
| $V_z/F$ | Apparent volume of distribution |
| $V_T$ | Volume of distribution |
| WHO | World Health Organisation |

# 2 Signatures

The following persons have read and agreed the content of this Statistical Analysis Plan:



#### 3 Introduction

This statistical analysis plan (SAP) is based on the current trial protocol (version 2, 23 January 2023). Where statistical methods differ substantially between this SAP and the protocol, that will be identified in this document.

This SAP describes the datasets and the statistical methods to be used for the reporting and analysis of all data collected during the trial except the PET data analysis which will be analysed and reported separately by Inviero.

If a future protocol amendment necessitates a substantial change to the statistical analysis of the trial data, this SAP will be amended accordingly. If, after database lock, additional analyses are required to supplement the planned analyses described in this SAP, those unplanned analyses will not be described in an amended SAP, but they will be identified in the integrated clinical study report (CSR). Any deviations from this SAP will be documented in the CSR.

This SAP has been written in consideration of the following guidelines:

- International Conference on Harmonization (ICH) E9, Guidance for Industry: Statistical Principles for Clinical Trials (ICH E9 1998)<sup>1</sup>; and
- ICH E3, Guidance for Industry: Structure and Content of Clinical Study Reports (ICH E3 1995)<sup>2</sup>.

Pharmacokinetic (PK) analysis will be done using WinNonlin v8.1 or higher on a Windows PC. Statistical analysis will be done using SAS <sup>®</sup> 9.4 or higher on a Windows PC.

# 4 Study objective(s) and endpoint(s)

# 4.1 Study objective(s)

## 4.1.1 Primary objective(s)

- To assess the pharmacodynamic (PD) response in peripheral blood mononuclear cells (PBMCs) following single and repeated oral doses of ASN51 in healthy subjects.
- To assess brain O-GlcNAcase occupancy using [18F]-IMA601 positron emission tomography (PET), following repeated oral doses of ASN51 in healthy subjects.

#### 4.1.2 Secondary objective(s)

- To assess the safety and tolerability of repeated oral doses of ASN51 in healthy subjects
- To assess the relationship between the plasma concentration of ASN51 and the time-course of brain O-GlcNAcase occupancy using [<sup>18</sup>F]-IMA601 PET, following repeated oral doses of ASN51 in healthy subjects

- To assess the pharmacokinetics (PK) of repeated doses of ASN51 in healthy subjects
- To assess the trough O-GlcNAcase occupancy of ASN51 after repeated doses in healthy subjects
- To determine the effect of food on the PD response in PBMCs following repeated ASN51 dosing in healthy subjects

## 4.2 Study endpoint(s)

## 4.2.1 Primary endpoint(s)

#### PD:

- Protein O-GlcNAcylation in PBMCs
- [18F]-IMA601 regional total volume of distribution (V<sub>T</sub>) at each brain scan

## 4.2.2 Secondary endpoint(s)

#### Safety and tolerability:

• vital signs (blood pressure, pulse rate, tympanic temperature, and respiratory rate), 12-lead safety electrocardiogram (ECG), physical and neurological examination, laboratory safety tests (haematology, clinical chemistry, coagulation, and urinalysis), Columbia-Suicide Severity Rating Scale (C-SSRS), and adverse events (AEs)

#### PK:

- plasma concentration of ASN51 at the time of each postdose PET scan
- PK parameters including C<sub>max</sub>, C<sub>max</sub>/Dose, t<sub>max</sub>, t½, λ<sub>Z</sub>, AUC<sub>tau</sub>, AUC<sub>last</sub>, AUC<sub>inf</sub>, AUC<sub>inf</sub> /Dose, %AUC<sub>extrap</sub>, CL<sub>SS</sub>/F, V<sub>Z</sub>/F, C<sub>trough</sub>, R<sub>ac(Cmax)</sub>, R<sub>ac(AUC)</sub>.

#### PD:

- Protein O-GlcNAcylation in PBMCs with or without prior feeding
- Trough [ $^{18}$ F]-IMA601 V<sub>T</sub>

#### PK/PD:

• relationship between ASN51 plasma concentration, PBMC target engagement, and brain receptor occupancy (RO) over time

## 4.3 Statistical hypotheses

The trial is an exploratory one, and there are no null hypotheses to be tested.

## 5 Study design

This is a phase 1, open-label, dose escalation, PET study to investigate the brain occupancy of O-GlcNAcase, and the PD response in PBMCs, after repeated doses of ASN51 in healthy subjects.

Enrolment of up to 12 healthy subjects is planned, in up to 2 groups (Groups 1 and 2). Each group will consist of up to 6 subjects.

All subjects will receive once-daily (QD) doses of ASN51, by mouth, for 14 days: Group 1 will receive ASN51 QD and Group 2 will receive ASN51 QD. Group 2 will proceed only if the safety and tolerability of the previous dose level are acceptable, and the plasma concentrations of ASN51 are predicted to remain below the toxicokinetic limit, as determined by the Safety Review Group (SRG; see protocol section 8.5).

On Day 11, to evaluate the effect of food on PBMC response, subjects will receive ASN51 in the fed state following a United States Food and Drug Administration (FDA) high-fat breakfast. Subject fasting requirements are further detailed in protocol section 11.

In each group, 2 subjects will have a PBMC-only study design (section 5.1.1) and 4 will have a PBMC and PET scanning study design (section 5.1.2).

Schematic diagrams of each study design are in protocol section 8.2.

#### **5.1.1 PBMC-only subjects**

2 subjects in each of Groups 1 and 2 will not have PET scans during the study. They will:

- be screened within 28 days before their first dose of trial medication.
- be resident on ward from 1 day before their first dose (Day –1) until 6 days after their final dose (Day 20).
- return for a follow-up visit 9–11 days after their final dose of trial medication (Days 23–25).

#### 5.1.2 PET subjects

4 subjects in each of Groups 1 and 2 will have PET scans during the study. PET subjects will:

- be screened within 21 days before imaging session 1 (see below).
- be resident on ward from 1 day before their first dose (Day -1) until 6 days after their final dose (Day 20); and have imaging sessions as described below.
- return for a follow-up visit 9–11 days after their final dose of trial medication (Day  $23 \pm 2$  days), or 2–4 days after imaging session 3 (see below), whichever is later.

PET subjects will have up to 3 imaging sessions, as follows.

- *Imaging session 1*. Subjects will have a baseline PET scan between Day –7 and Day –3. Subjects will be admitted to the ward the day before their baseline PET scan, and be discharged the following day after their scan.
- *Imaging session 2*. Subjects will have an on-treatment PET scan at about 5 h postdose on Day 1.
- *Imaging session 3*. Subjects will have an on-treatment PET scan at 3–9 days after their final dose of ASN51:
  - 3 subjects per group on Day 17
  - 1 subject on Day 22 (± 1 day) (Group 1 only)
  - 1 subject on Day 23 ( $\pm$  1 day) (Group 2 only)

The timing of on-treatment PET scans (imaging sessions 2 and 3) may be altered based on emerging data or study logistical requirements.

Subjects will receive an intravenous (IV) dose of the radiolabelled tracer, [18F]-IMA601, at the start of each PET scan.

Arterial blood sampling will be done during each PET scan to quantify the parent tracer-related radioactivity over the course of the PET scan, and to establish a tracer metabolite-corrected plasma input function. The total arterial blood volume required for each tracer injection will not exceed 120 mL. Arterial cannulation and arterial blood sampling may be reduced or removed if analysis of PET data from previous subjects indicates that non-invasive analysis of the PET scan data can be done. If a non-invasive analysis is not possible, the use of an arterial cannula with each PET scan will continue through the study.

In the case of a technical failure (such as unsuccessful tracer synthesis), subjects may be asked to attend an additional on-treatment imaging session as described in section 12.2 of the protocol. However, no subject will have more than 3 PET scans and 3 doses of [<sup>18</sup>F]-IMA601 during the study. See section 8.2 of the protocol for the design flow charts.

#### 6 Time and events table

Please refer to section 12.1 of the protocol, version 2, dated 23 January 2023 and file note Ward 2.

# 7 Planned analyses

No interim analyses are planned. However, data will be reviewed for dose selection.

## 7.1 Interim analyses

No interim analyses are planned. However, safety and pharmacokinetic data from Group 1 will be reviewed before proceeding to Group 2.

## 7.2 Final analysis

The database will be locked once all subjects have completed the study, data have been entered, and queries resolved. The final analysis will be carried out following database lock.

#### 7.2.1 Persons responsible for analysis

Statistician

## 8 Sample size considerations

## 8.1 Sample size assumptions

Since this trial is hypothesis generating, no formal calculation of sample size is appropriate.

The sample size chosen is considered adequate to allow modelling of the relationship between ASN51 plasma concentrations and pharmacodynamic target engagement using an exploratory PBMC protein O-GlcNAcylation assay.

PET analyses of 8 subjects is sufficient to define the occupancy of O-GlcNAcase and is within the range generally accepted for PET studies.

# 9 Analysis populations

The following populations will be identified:

Safety population: All subjects who received at least one dose of study drug

PET population: All subjects in the safety population who had a baseline PET

scan, at least 1 post-baseline PET scan, and a PK result

immediately preceding a PET scan

PD analysis population: All subjects in the safety population for who a PBMC measure

is available.

PK analysis population: The PK analysis population will consist of the subjects who

provide evaluable data for the comparisons of interest. These

subjects should have at least one quantifiable plasma concentration, should not have violated any major entry criterion likely to confound the PK analysis, and should not have deviated significantly from the protocol between

nave activated significantly from the protector of

enrolment and successful study completion

The primary endpoints will be analysed using the PET and PD populations. The secondary endpoints will be analysed using the Safety, PET and PD populations.

## 9.1 Analysis datasets

All analysis datasets will be based on observed data, except as outlined in Section 12.2.

## 10 Treatment comparisons

The treatment comparison of interest is study drug between ascending doses.

## 11 General considerations for data analyses

## 11.1 Data display treatment and other subgroup descriptors

The sort order for treatment groups will be study treatment in ascending dose order.

Listings of data will be sorted and displayed by treatment group, subject number, and also by date and time if applicable.

The treatment descriptions to be used on all tables and listings are:

#### **Treatment Groups**

ASN51 (QD for 14 Days) ASN51 (QD for 14 Days)

## 11.2 Conventions for summary statistics and data displays

The minimum set of summary statistics for numeric variables will be: n, mean, standard deviation, median, minimum, and maximum. 95% confidence intervals (CI) will be presented where appropriate for data interpretation.

Categorical data will be summarised in frequency tables with n and percentage. Summaries of a categorical variable will include all recorded values.

The minimum and maximum values will be presented with the same number of decimal places as the raw data collected on the CRF (or to 3 significant figures for derived parameters less than 100 and as integers for values more than 99). The mean and percentiles (eg median) will be presented using one additional decimal place. The standard deviation and standard error will be presented using two additional decimal places.

# 12 Data handling conventions

# 12.1 Premature withdrawal and missing data

All subjects who withdraw prematurely from the study or study drug will be included in the statistical analyses.

If a subject completes the treatment period but has missing data, then this will be made apparent in the subject listings. Missing data will not be imputed except for as outlined in Section 12.2.

If the study is prematurely discontinued, all available data will be listed and a review will be carried out to assess which statistical analyses are still considered appropriate.

Data collected at unscheduled time points during the study will not be used in the summaries or data analyses. They will be included in the listings.

If time information (ie hours and/or minutes) for adverse events (AEs) or concomitant medication is missing, but the day is present, then the time will be calculated in days. If date information is partial or missing, then any derived times (eg AE start time from last study medication) will be listed as missing.

Conventions for handling missing plasma concentrations are given in Appendix B: Pharmacokinetic analysis

#### 12.2 Derived and transformed data

Baseline will be considered to be the latest value obtained before study drug administration (eg Day 1, pre-dose; or Day –1 if not recorded at pre-dose; or screening if not recorded at pre-dose or on Day –1).

Laboratory data will be reported in standard units. Out-of-range laboratory tests may be repeated. If a test is out of-range at baseline and repeated before dosing, the latest repeat value before dosing will be used as baseline. However, if a test is out-of-range and repeated at any other time during the study, the out-of-range value (not the repeat value) will be included in statistical summaries.

Triplicate ECG and vital sign measurements will be made at screening and the mean of the three measurements for each subject will be used for analysis.

Triplicate PBMC measurements will be made and the mean of the three measurements for each subject will be used for analysis.

The PK parameters to be derived are given in Appendix B: Pharmacokinetic analysis.

#### 12.3 Assessment windows

No assessment windows are defined for this report.

## 12.4 Vital signs reference ranges

The following vital signs ranges will be used:

| Vital Sign | Range |
|---------------------------------|-------------------|
| Seated systolic blood pressure | 90–140 mm Hg |
| Seated diastolic blood pressure | 40–90 mm Hg |
| Seated pulse rate | 40–100 beats/min |
| Tympanic temperature | 35.5–37.8°C |
| Respiratory rate | 10–16 breaths/min |

## 13 Study population

## 13.1 Disposition of subjects

The disposition of all subjects in all populations will be summarised including: number of subjects by treatment; number completing the study, by treatment; and number withdrawn from the study. Screen failures will also be listed and summarised.

All subjects who withdraw or are withdrawn from the study will be listed, by treatment, with the reason for withdrawal.

A listing of analysis populations will be provided.

#### 13.2 Protocol deviations

Before closing the database, data listings will be reviewed to identify any significant deviations and determine whether the data should be excluded from any analysis populations.

Major protocol deviations include subjects who:

- Entered the study even though they did not satisfy the entry criteria.
- Met the criteria for withdrawal from the study but were not withdrawn.
- Received the wrong treatment or incorrect dose.
- Received an excluded concomitant therapy.
- Received investigational product(s) past the expiration date.

In addition, subjects with minor time deviations (measurements taken outside the allowable windows) will be identified. Allowable time windows for pharmacokinetic samples and other procedures are given in 12.2 of the study protocol.

## 13.3 Demographic and baseline characteristics

Demographic and baseline characteristics (eg physical examination, vital signs and ECGs) will be listed and summarised.

Subjects who take concomitant medication will be listed. All non-trial medication will be coded using the latest version of the World Health Organisation (WHO) ATC index (version 2021 or higher).

Medical and surgical history data will also be listed. Medical and surgical history will be coded using the version of the Medical Dictionary for Regulatory Activities (MedDRA) current at the time of database lock.

## 13.4 Treatment compliance

Dates and times of dosing will be listed.

## 14 Safety analyses

Summaries and listings of safety data will use the safety population.

## 14.1 Extent of exposure

The dates and times of treatment dosing will be listed to indicate exposure to the study medication.

#### 14.2 Adverse events

AEs will be coded using the version of the Medical Dictionary for Regulatory Activities (MedDRA) which is current at the time of database lock (version 25.1 or higher).

All AEs will be listed.

The number of subjects with at least one treatment-emergent adverse event (TEAE) per treatment will be tabulated by actual treatment and MedDRA system organ class. A TEAE is defined as an event emerging during treatment (having been absent pre-treatment) or that worsens after treatment<sup>1</sup>.

For each of the following, the number of TEAEs and the number of subjects with TEAEs will be summarised by treatment:

- TEAEs, by system organ class and preferred term
- Drug-related ("possibly", "probably" or "definitely" as recorded by the investigator) TEAEs, by system organ class and preferred term

Subjects with more than one TEAE will be counted only once, at the greatest severity or causality, for each system organ class/preferred term. Multiple TEAEs in a subject will be counted once per system organ class and preferred term. AEs with missing severity and/or causality will be treated as severe and definitely related, respectively.

Summaries will be sorted by system organ class and decreasing total incidence of preferred term.

# 14.3 Deaths, serious adverse events and other significant adverse events

Deaths and serious adverse events (SAEs) will be listed separately (fatal events separate from non-fatal events). Other significant AEs, as identified by the investigator in the CRF, will be listed separately.

## 14.4 Adverse events leading to withdrawal from the study

AEs leading to withdrawal will be listed separately.

## 14.5 Clinical laboratory evaluations

Data from haematology, coagulation, urinalysis, and clinical chemistry will be summarised by treatment.

The laboratory tests with normal ranges that are different from the ranges most commonly used in the study (reference ranges) are listed in Appendix A: Laboratory tests with different ranges.

Data from haematology, coagulation, and clinical chemistry outside the normal ranges (used to assign clinical significance) and/or reference ranges (the most commonly used in the study) will be listed. Data outside the reference ranges will be summarised.

## 14.6 Other safety measures

#### 14.6.1 Vital signs

Vital signs evaluation at each planned assessment, and change in vital signs from baseline (Day 1, pre-dose) at each planned post baseline assessment, will be summarised by actual treatment.

Vital signs data outside of the normal range will be listed and summarised.

A separate listing of vital sign findings, classified as clinically significant by the investigator will also be provided.

#### 14.6.2 ECG

QT interval data will be presented using Fridericia's (QTcF) corrections.

ECG variables will be summarised by treatment and time point. Differences from baseline (Day 1 pre-dose) will be summarised by treatment and time point.

QTcF values > 450 msec, PR interval shortening < 110 msec, and PR interval prolongation >220 msec, and increases of QTcF from baseline of > 30 msec and > 60 msec, will be listed by treatment and timepoint and summarised. A separate listing of ECG findings classified as abnormal by the investigator will also be provided.

#### 14.6.3 Physical examination

Abnormal physical and neurological examination findings will be listed.

#### 14.6.4 Columbia-Suicide Severity Rating Scale (C-SSRS)

Positive C-SSRS data will be listed.

## 15 Pharmacokinetic analyses

The PK parameters to be derived are given in Appendix B: Pharmacokinetic analysis.

PK concentration data will be summarised using the PK analysis population.

Plasma concentrations and PK parameters will be listed and summarised, by treatment, using descriptive statistics. Individual and mean plasma concentration—time profiles will be presented graphically. All available data will be used to derive PK parameters in individual subjects.

For log-transformed parameters, the primary measure of central tendency will be the geometric mean<sup>4</sup>; for other parameters, it will be the arithmetic mean or median.

For all variables, N (number of subjects receiving the treatment/formulation in the population), n (number of observations), arithmetic mean, median, minimum, maximum, standard deviation (SD), %CV, and the 95% CI for the arithmetic mean will be provided. For log-transformed variables, all of the above plus the geometric mean, which is the anti-logged arithmetic mean of log-transformed variables, its 95% CI and the SD of the logs will be provided.

The between-subject CV will be calculated using:

- 1. %CVb = 100 \* (SD/mean) with SD and mean of untransformed data
- 2. %CVb =  $100 * \sqrt{(\exp(SD)^2 1)}$  with SD of log-transformed data

#### 15.1 Pharmacokinetic concentration data

Plasma concentrations will be listed and summarised by treatment.

Using actual sample times, linear and semi-logarithmic concentration-time plots will be prepared by treatment and synoptic linear and semi-logarithmic plasma concentration-time plots of ASN51 will be prepared for each Day. In addition to the plots of concentrations on PK days, separate plots of trough concentrations for ASN51 will be prepared. The same linear and logarithmic scales will be used for each subject. The linear and semi-logarithmic plots for a given treatment will be presented on the same page.

Nominal blood sampling times will be used to calculate the mean (SD) drug concentrations at each time point.

Mean(+/- SD), and spaghetti plasma concentration versus time plots will be presented for ASN51 per treatment (synoptic plot) (normal scale and log-linear scale).

## 15.2 Pharmacokinetic parameters

The pharmacokinetic parameters will be listed and summarised by treatment.

## 16 Pharmacodynamic analyses

Protein O-GlcNAcylation in PBMCs at each planned assessment, and change in protein O-GlcNAcylation in PBMCs from baseline (Day 1, pre-dose) at each planned post baseline assessment, will be summarised by actual treatment using the PD population.

Time invariance of target engagement will be investigated by comparing the PD and PK/PD relationship over time.

Food effect on the PBMC assay will be investigated by comparing Day 11 and 14 PBMC data descriptively.

In addition to the descriptive statistics of the PBMC data (ie N, mean, median, SD, min, max, CV%), time-matched change from baseline PBMC parameters (Day 1 vs Day 14, and Day 11 vs Day 14) will be assessed using an Analyses of variance (ANOVA) approach. ANOVA will be performed on the natural log(ln)-transformed PBMC parameters. Each ANOVA will include calculation of least square means (LSM), the difference between LSM of the two conditions, and the standard error and 90% confidence interval (CI) associated with this difference. The LSM, difference in LSMs, and associated 90% CI will be back transformed to present geometric LSM, the ratio of geometric means, and associated 90% CI. The 90% CI of geometric mean ratio will be calculated to check whether it lies within the interval 0.70 to 1.43.

Furthermore, PBMC data and plasma concentration data of Day 1 and Day 14 will be investigated by a regression analysis, where the slopes and intercepts will be compared statistically for each treatment. The change from baseline of PMBC data will be analysed using analysis of covariance (ANCOVA). Time point, PK concentration and PK concentration by time point interaction will be fitted as fixed effects. PK concentration will be treated as a continuous covariate and time point will be fitted as a categorical covariate. The estimates, standard errors, associated 95% CI and P-values will be reported.

# 17 Changes from the protocol specified statistical analysis

After the study was submitted to the MHRA and ethics committee the following changes were made to the analyses:

• Various updates to scheduled timepoints have been made as document in file note ward 2.

#### 18 References

- 1. International Conference on Harmonization, 1998. Statistical Principles for Clinical Trials ICH Harmonised Tripartite Guideline. Guidance for Industry, E9, FDA federal register, Vol 63, 1998, p49583. Available at: http://www.fda.gov/cder/guidance.
- 2. International Conference on Harmonization, 1995. Structure and Content of Clinical Study Reports ICH Harmonised Tripartite Guideline. Guidance for Industry, E3, FDA federal register, Vol 61, 1996, p37320. Available at: http://www.fda.gov/cder/guidance.
- 3. International Conference on Harmonisation, 2005. Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs. Concept paper, Guidance for Industry, E14, Center for Drug Evaluation and Research (CDER). Available at: http://www.fda.gov/cder/guidance/6922fnl.htm.
- 4. Julious, SA & Debarnot, CAM (2000) "Why are Pharmacokinetic Data Summarised by Arithmetic Means?", Journal of Biopharmaceutical Statistics, 10 (1), p55-71

#### 19 ATTACHMENTS

## 19.1 Table of contents for data display specifications

For overall page layout refer to Appendix C: Sample page.

The numbering in the tables below will take precedence over the numbering in the shells.

The following tables and figures will be produced (templates provided in Sections 19.2.1 and 19.2.2):

| Table | Description | Population | Source<br>Listing | Template<br>(Shells below) |
|---|---|---|---|---|
| 10.1 | Summary of subject disposition | Safety | 16.2.1.2 | T SD1 |
| | | | 16.2.1.3 | |
| | | | 16.2.3.1 | |
| 14.1 | DEMOGRAPHIC DATA | | | |
| 14.1 | Summary of demographic characteristics | Safety | 16.2.4.1 | <u>T DM1</u> |
| 14.2 | PHARMACOKINETIC AND PHARMACODYNAMIC DATA | | | |
| 14.2.1.1 | Summary of ASN51 plasma pharmacokinetic concentration-time data [units] | PK analysis | 16.2.6.1.1 | <u>T_PK1</u> |
| 14.2.1.2 | Summary of derived ASN51 plasma pharmacokinetic parameters | PK analysis | 16.2.6.1.2 | T PK3 |
| | | | 16.2.6.1.3 | |
| 14.2.1.3 | Summary of log-transformed derived ASN51 plasma pharmacokinetic | PK analysis | 16.2.6.1.2 | <u>T_PK4</u> |
| | parameters | | 16.2.6.1.3 | |
| 14.2.2.1 | Summary of plasma PBMC data (% above baseline) | PD analysis | 16.2.6.2 | <u>T_VS1</u> |
| 14.2.2.2 | Summary of analysis of time-matched change from baseline plasma | PD analysis | 16.2.6.2 | T_ANOVA1 |
| | PBMC data using analysis of variance (Day 1 vs Day 14 and Day 11 vs Day 14) | | | |
| 14.2.2.3 | Summary of ANCOVA analysis of PBMC and PK concentration to compare intercepts and slopes between Day 1 and Day 14 | PD analysis | 16.2.6.2 | T REGR |
| 14.3 | SAFETY DATA | | | |
| 14.3.1.1 | Overall summary of treatment-emergent adverse events | Safety | 16.2.7.1 | T_AE2 |
| 14.3.1.2 | Summary of treatment-emergent adverse events | Safety | 16.2.7.1 | <u>T AE1</u> |
| 14.3.1.3 | Summary of drug-related treatment-emergent adverse events | Safety | 16.2.7.1 | <u>T_AE1</u> |
| 14.3.2.1 | Listing of fatal adverse events | Safety | 16.2.7.1 | L AE1 PG |
| 14.3.2.2 | Listing of non-fatal serious adverse events | Safety | 16.2.7.1 | L AE1 PG |
| 14.3.2.3 | Listing of other significant adverse events | Safety | 16.2.7.1 | L_AE1_PG |
| 14.3.3 | Narratives of deaths, other serious and significant adverse events | Safety | | - |
| 14.3.4.1 | Summary of laboratory values outside the reference range by treatment | Safety | 16.2.8.1 | <u>T_LB1</u> |
| | and planned relative time | | 16.2.8.2 | |
| | | | 16.2.8.3 | |

13 June 2023 

| Table | Description | Population | Source<br>Listing | Template<br>(Shells below) |
|---|---|---|---|---|
| 14.3.4.2 | Summary of laboratory values outside the reference range by treatment | Safety | 16.2.8.1<br>16.2.8.2<br>16.2.8.3 | T_LB3 |
| 14.3.5.1 | Summary of chemistry laboratory values | Safety | 16.4 | T LB2 |
| 14.3.5.2 | Summary of haematology laboratory values | Safety | 16.4 | T LB2 |
| 14.3.5.3 | Summary of coagulation laboratory values | Safety | 16.4 | T LB2 |
| 14.3.5.4 | Summary of urinalysis results | Safety | 16.4 | T UR1 |
| 14.3.6.1 | Summary of vital signs | Safety | 16.4 | T VS1 |
| 14.3.6.2 | Summary of vital signs outside the normal range by treatment, planned relative time and parameter | Safety | 16.2.9.1 | <u>T_VS2</u> |
| 14.3.6.3 | Summary of vital signs outside the normal range by treatment and parameter (excluding baseline time point) | Safety | 16.2.9.1 | <u>T_VS3</u> |
| 14.3.7.1 | Summary of ECG values | Safety | 16.4 | T EG2 |
| 14.3.7.2 | Summary of QTcF and PR interval values outside the normal range by treatment, planned relative time and category | Safety | 16.2.9.3 | T_EG3 |
| 14.3.7.3 | Summary of QTcF and PR interval values outside the normal range by treatment and category | Safety | 16.2.9.3 | T_EG4 |

| Figure | Description | Population | Source<br>Listing | Template<br>(Shells below) |
|---|---|---|---|---|
| 14.2 | PHARMACOKINETIC AND PHARMACODYNAMIC DATA | | | |
| 14.2.1 | Individual ASN51 plasma concentration-time plots (linear and semi-log) | PK analysis | 16.2.6.1.1 | F_PK1 |
| 14.2.2 | Mean (+/- SD) ASN51 plasma concentration-time plots (linear and semi-log) | PK analysis | 16.2.6.1.1 | <u>F_PK2</u> |
| 14.2.3 | Mean ASN51 plasma concentration-time plots (linear and semi-log) | PK analysis | 16.2.6.1.1 | F PK2 |
| 14.2.4 | Individual ASN51 plasma pre-dose concentration versus day | PK analysis | 16.2.6.1.1 | F_PK5 |
| 14.2.5 | Mean (+/- SD) ASN51 plasma pre-dose concentration versus day | PK analysis | 16.2.6.1.1 | <u>F_PK6</u> |

13 June 2023 

| Figure | Description | Population | Source<br>Listing | Template<br>(Shells below) |
|---|---|---|---|---|
| 14.3 | SAFETY DATA | | | |
| 14.3.1 | Individual systolic blood pressure-time plots | Safety | 16.4 | F SAF1 |
| 14.3.2 | Individual diastolic blood pressure-time plots | Safety | 16.4 | F SAF1 |
| 14.3.3 | Individual heart rate-time plots | Safety | 16.4 | F SAF1 |
| 14.3.4 | Individual QTcF-time plots | Safety | 16.4 | F SAF1 |

The following abbreviated listings will be produced (templates provided in Section 19.2.3):

| Listing | Description | Template (Shells<br>below) |
|---|---|---|
| 16.2.1 | Study dates & disposition of subjects | |
| 16.2.1.1 | Listing of study dates | L SD1 PG |
| 16.2.1.2 | Listing of reasons for withdrawal | L SD2 PG |
| 16.2.1.3 | Listing of subjects screened but not enrolled | L SD3 PG |
| 16.2.2 | Protocol deviations | |
| 16.2.2.1 | Listing of subjects with inclusion/exclusion criteria deviations | L DV1 PG |
| 16.2.2.2 | Listing of subjects with time deviations | L TD1 PG |
| 16.2.2.3 | Listing of subjects with other protocol deviations | L DV2 PG |
| 16.2.3 | Analysis sets, including subjects excluded from analysis | |
| 16.2.3.1 | Listing of analysis populations | L AN1 PG |
| 16.2.4 | Demographic data & concomitant medication | |
| 16.2.4.1 | Listing of demographic characteristics | L DM1 PG |
| 16.2.4.2 | Listing of concomitant medications | L CM1 PG |
| 16.2.4.3 | Listing of medical history | L MH1 X |
| 16.2.5 | Study drug administration | |
| 16.2.5.1 | Listing of exposure data | L EX1 PG |
| 16.2.6 | Pharmacokinetic and pharmacodynamic data | |
| 16.2.6.1.1 | Listing of ASN51 plasma pharmacokinetic concentration-time data | L PK1 PG |

13 June 2023 

| Listing | Description | Template (Shells |
|---|---|---|
| | | below) |
| 16.2.6.1.2 | Listing of derived ASN51 plasma pharmacokinetic parameters | L PK4 PG |
| 16.2.6.1.3 | Listing of derived ASN51 Ctrough (ng/mL) pharmacokinetic parameter | L PK4 PG |
| 16.2.6.1.4 | Individual ASN51 plasma concentration-time plots for estimation of $\lambda z$ , with regression line | <u>F_PK10</u> |
| 16.2.6.2 | Listing of plasma PBMC data | L_PBMC_PG |
| 16.2.7 | Adverse events | |
| 16.2.7.1 | Listing of all adverse events | L AE1 PG |
| 16.2.7.2 | Listing of serious adverse events | L AE1 PG |
| 16.2.7.3 | Listing of adverse events leading to withdrawal from study | L AE1 PG |
| 16.2.8 | Laboratory values | |
| 16.2.8.1 | Listing of clinical chemistry data outside the normal range | L LB1 PG |
| 16.2.8.2 | Listing of haematology data outside the normal range | L LB1 PG |
| 16.2.8.3 | Listing of coagulation data outside the normal range | L LB1 PG |
| 16.2.9 | Vital signs, ECG variables, physical and neurological findings and | |
| 16201 | C-SSRS | T TICL DC |
| 16.2.9.1 | Listing of vital signs outside the normal range | L_VS1_PG |
| 16.2.9.2 | Listing of clinically significant vital signs | L VS2 PG |
| 16.2.9.3 | Listing of QTcF and PR interval values outside the normal range | <u>L EG1 PG</u> |
| 16.2.9.4 | Listing of abnormal ECG findings | L EG2 PG |
| 16.2.9.5 | Listing of abnormal physical examination findings | L PE1 PG |
| 16.2.9.6 | Listing of abnormal neurological examination findings | L NEURO PG |
| 16.2.9.7 | Listing of positive Columbia-Suicide Severity Rating Scale data | L CSS PG |

<sup>\*</sup> ICH does not require full listings of lab data so only subjects with out-of-range values will be listed.

Complete listings of all data collected in this study will also be produced.

# 19.2 Data Display Specifications

Footnote "Note: Subjects received ASN51 in the fed state on Day 11 only" will be added to any outputs with Day 11

## **19.2.1** Table Outlines

#### Template T\_SD1

Table 10.1 Summary of subject disposition

| | | | Treatment 1 | Treatment 2 | |
|---|---|---|---|---|---|
| Characteristics | Status | Reason for Withdrawal | (N=xx) | (N=xx) | All Subjects |
| | | | n (%) | n (%) | n (%) |
| Screened population | Total | | | | XX |
| | Included | | | | XX |
| | Excluded | Not satisfying | | | XX |
| | | inclusion/exclusion criteria | | | |
| | | Declined to participate | | | XX |
| | | Other | | | XX |
| Safety population | Included | | XX | XX | XX |
| | Completed | | xx (xx) | xx (xx) | xx (xx) |
| | Withdrawn | | xx (xx) | xx (xx) | xx (xx) |
| | | Death | xx (xx) | xx (xx) | xx (xx) |
| | | Adverse Events | xx (xx) | xx (xx) | xx (xx) |
| | | Withdrawal by subject | xx (xx) | xx (xx) | xx (xx) |
| | | Study terminated by Sponsor | xx (xx) | xx (xx) | xx (xx) |
| | | Lost to follow-up | xx (xx) | xx (xx) | xx(xx) |
| | | Other | xx (xx) | xx (xx) | xx (xx) |
| Alternative 1 (if applicable) | Included | | | | |
| Alternative 2 (if applicable) | Included | | | | |

Source: Listing 16.2.xx

Note: Subjects received ASN51 in the fed state on Day 11 only

Programming notes: Continued with all treatment groups

13 June 2023 

#### Template T\_DM1

Table 14.1 Summary of demographic characteristics

| Variable | Statistics | Treatment 1(N=xx) | Treatment 2<br>(N=xx) | All Subjects (N=xx) |
|---|---|---|---|---|
| Age (y) | n | | | |
| | Mean | | | |
| | SD | | | |
| | Median | | | |
| | Min | | | |
| | Max | | | |
| Sex (%) | Female | | | |
| | Male | | | |
| Race (%) | American Indian or Alaskan | | | |
| | Native | | | |
| | Asian | | | |
| | Black | | | |
| | Native Hawaiian or other | | | |
| | Pacific Islander | | | |
| | White | | | |
| | Other | | | |
| Ethnicity (%) | Hispanic or Latino | | | |
| | Not Hispanic or Latino | | | |
| Height (cm) | n | | | |
| | Mean | | | |
| | SD | | | |
| | Median | | | |
| | Min | | | |
| | Max | | | |
| Weight (kg) | n | | | |
| | Mean | | | |
| | SD | | | |
| | Median | | | |
| | Min | | | |

13 June 2023 

| Variable | Statistics | Treatment 1 | Treatment 2 | All Subjects (N=xx) |
|--------------|------------|-------------|-------------|---------------------|
| | - | (N=xx) | (N=xx) | <del>-</del> |
| | Max | | | |
| BMI (kg/m2) | n | | | |
| | Mean | | | |
| | SD | | | |
| | Median | | | |
| | Min | | | |
| | Max | | | |
| Smoking | Never | | | |
| History (%) | Former | | | |
| | Current | | | |
| Cigarettes* | n | | | |
| (daily) | Mean | | | |
| | SD | | | |
| | Median | | | |
| | Min | | | |
| | Max | | | |
| Alcohol* | n | | | |
| (units/week) | Mean | | | |
| | SD | | | |
| | Median | | | |
| | Min | | | |
| | Max | | | |

Source: Listing 16.2.xx

<sup>\*</sup>includes only those subjects who smoke/drink alcohol

#### Template T\_PK1

Table 14..2.xx Summary of ASN51 plasma pharmacokinetic concentration-time data [units]

| Treatment | Planned<br>Relative<br>Time | n | No.<br>Imputed | Mean | 95% CI<br>(Lower,Upper) | SD | %CVb | Median | Min | Max |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment 1 | Pre-dose | х | х | XXXX.X | (xxxx.x,xxxx.x) | | XX.X | xxxx.x | XXXX | XXXX |
| (N=xx) | 30 min | х | х | XXXX.X | (xxxx.x,xxxx.x) | XX.XX | XX.X | xxxx.x | XXXX | XXXX |
| | 1 h | х | X | XXXX.X | (xxxx.x,xxxx.x) | xx.xx | XX.X | XXXX.X | XXXX | XXXX |
| Treatment 2 | Pre-dose | х | x | xxxx.x | (xxxx.x,xxxx.x) | xx.xx | xx.x | xxxx.x | XXXX | XXXX |
| (N=xx) | 30 min | х | x | XXXX.X | (xxxx.x,xxxx.x) | xx.xx | XX.X | xxxx.x | xxxx | XXXX |
| | 1 h | х | x | XXXX.X | (xxxx.x,xxxx.x) | XX.XX | XX.X | xxxx.x | XXXX | XXXX |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels and timepoints

Column "No. Imputed" is not required for summary of PBMC data

#### Template T\_PK3

Table 14..2.xx Summary of derived ASN51 plasma pharmacokinetic parameters

| | | | | | 95% CI | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Parameter | Treatment | Study Day | n | Mean | (Lower,Upper) | SD | %CVb | Median | Min | Max |
| AUC <sub>t</sub> (units) | Treatment 1 (N=xx) | | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | XX.X | XXXX.XX | xxxx.x | xxxx.x |
| | Treatment 2 (N=xx) | | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | XX.X | XXXX.XX | xxxx.x | xxxx.x |
| C <sub>max</sub> (units) | Treatment 1 (N=xx) | | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | XX.X | XXXX.XX | xxxx.x | xxxx.x |
| | Treatment 2 (N=xx) | | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | XX.X | XXXX.XX | xxxx.x | xxxx.x |

Source: Listing 16.2.xx

 $R_{ac}$  (AUC) =  $R_{ac}$  (AUC<sub>tau</sub>) Day 14 /  $R_{ac}$ (AUC<sub>tau</sub>) Day 1  $R_{ac}$  (C<sub>max</sub>) =  $R_{ac}$  (C<sub>max</sub>) Day 14/ $R_{ac}$ (C<sub>max</sub>) Day 1

Programming notes: Continued with all dose levels, timepoints and parameters

13 June 2023 

#### Template T\_PK4

Table 14..2.xx Summary of log-transformed derived ASN51 plasma pharmacokinetic parameters {by group}

| Parameter | Treatment | Study Day | n | Geom<br>Mean | 95% Cl<br>(Lower,Upper) | SD (logs) | %CVb |
|---|---|---|---|---|---|---|---|
| AUC <sub>last</sub> (units) | Treatment 1 (N=xx) | х | Х | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XXX | xx.xx |
| | Treatment 2 (N=xx) | х | Х | XXXX.XX | (xxxx.xx,xxxx.xx) | xx.xxx | xx.xx |
| C <sub>max</sub> (units) | Treatment 1 (N=xx) | x | Х | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | xx.xx |
| | Treatment 2 (N=xx) | X | Х | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | xx.xx |

Source: Listing 16.2.xx

Programming notes: Continued with all dose levels, timepoints and parameters

#### Template T\_ANOVA1

Table 14.2.xx Summary of analysis of time-matched change from baseline plasma PBMC data using analysis of variance -Day 1 vs Day 14 and Day 11 vs Day 14 (% above baseline)

| | LS | | | S Means Day 1 vs | | | y 14 | Day | ay 14 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Planned<br>RelativeTime | Day 1 | Day 1 Day 11 | | Geometric<br>Mean Ratio | SE | 90% CI | Geometric<br>Mean Ratio | SE | 90% CI |
| Treatment 1 (N=xx) | Pre-dose | NA | XXXX | XXXX | NA | NA | NA | x.xx | x.xx | x.xx |
| | 8 h | XXXXX | XXXX | XXXX | x.xx | x.xx | (x.xx, x.xx) | x.xx | x.xx | (x.xx, x.xx) |
| | 12 h | XXXXX | XXXX | XXXX | x.xx | x.xx | (x.xx, x.xx) | x.xx | x.xx | (x.xx, x.xx) |
| Treatment 2 (N=xx) | Pre-dose | NA | XXXX | XXXX | NA | NA | NA | x.xx | x.xx | x.xx |
| | 8 h | XXXXX | XXXX | XXXX | x.xx | x.xx | (x.xx, x.xx) | x.xx | x.xx | (x.xx, x.xx) |
| | 12 h | XXXXX | XXXX | XXXX | x.xx | x.xx | (x.xx, x.xx) | x.xx | x.xx | (x.xx, x.xx) |

Source: Listing 16.2.xx

NA = not applicable

#### Template T\_REGR

Table 14.2.xx Summary of ANCOVA analysis of PBMC and PK concentration to compare intercepts and slopes between Day 1 and Day 14

| Treatment | <u>Parameter</u> | Estimate | SE | 95% CI | P-Value |
|---|---|---|---|---|---|
| Treatment 1 (N=xx) | Intercept | xx.x | XX.XX | x.xxx | X.XXX |
| | PK Concentration | xx.x | XX.XX | x.xxx | X.XXX |
| | Day 1 | xx.x | XX.XX | x.xxx | X.XXX |
| | Day 14 | XX.X | XX.XX | x.xxx | x.xxx |
| | PK Concentration*Day 1 | XX.X | XX.XX | x.xxx | x.xxx |
| | PK Concentration*Day 14 | XX.X | XX.XX | x.xxx | X.XXX |
| Treatment 2 (N=xx) | Intercept | xx.x | XX.XX | x.xxx | x.xxx |
| | PK Concentration | xx.x | XX.XX | x.xxx | X.XXX |
| | Day 1 | XX.X | XX.XX | x.xxx | x.xxx |
| | Day 14 | XX.X | XX.XX | x.xxx | x.xxx |
| | PK Concentration*Day 1 | xx.x | XX.XX | x.xxx | x.xxx |
| | PK Concentration*Day 14 | XX.X | XX.XX | X.XXX | X.XXX |

Source: Listing 16.2.xx

Programming notes: Include timepoints: 8 h, 12h and 24 h

13 June 2023 

#### Template T\_AE2

Table 14.3.3.xx Overall summary of treatment-emergent adverse events

| Number of Subjects with | Treatment 1 (N=xx)<br>n (%) | Treatment 1 (N=xx)<br>n (%) | All Subjects (N=xx)<br>n (%) |
|---|---|---|---|
| Any TEAE | x (xx.x) [xx] | x (xx.x) [xx] | x (xx.x) [xx] |
| Any serious TEAE | x (xx.x) [xx] | x (xx.x) [xx] | x (xx.x) [xx] |
| Any TEAE leading to withdrawal | x (xx.x) [xx] | x (xx.x) [xx] | x (xx.x) [xx] |
| Any drug-related TEAE | x (xx.x) [xx] | x (xx.x) [xx] | x (xx.x) [xx] |
| Any TEAE with mild as worst severity | x (xx.x) | x (xx.x) | x (xx.x) |
| Any TEAE with moderate as worst severity Any TEAE with severe as worst severity | | | |

Source: Listing 16.2.xx

n = number of subjects
[] = number of TEAEs

Programming notes: Continued with all treatment groups

13 June 2023 

#### Template T\_AE1

Table 14.3.3.xx Summary of treatment-emergent adverse events

| System Organ Class* Preferred Term | | Treatment 1 (N=xx)<br>n (%) | Treatment 2 (N=xx)<br>n (%) | All Subjects (N=xx)<br>n (%) |
|---|---|---|---|---|
| Number of subjects with TEAEs | | x (xx.x) | x (xx.x) | |
| Gastrointestinal disorders | Total number of subjects | x (xx.x) | x (xx.x) | |
| | Abdominal discomfort | x (xx.x) [xx] | x (xx.x) [xx] | |
| | Abdominal pain | x (xx.x) [xx] | x (xx.x) [xx] | |
| Nervous system disorders | Total number of subjects | | | |
| | Dizziness | | | |
| | Headache | | | |

Source: Listing 16.2.xx

n = number of subjects (subjects with >1 TEAE are counted only once per system organ class and preferred term)

[] = number of TEAEs

Programming notes: Continued with all treatment groups

SOCs and PTs are sorted in decreasing order of frequency

Presented for all applicable MedDRA system organ classes and terms.

13 June 2023 

<sup>\*</sup>Coded using MedDRA version xx.x

Template T\_LB1

Table 14.3.4.xx Summary of laboratory values outside the reference range by treatment and planned relative time

Laboratory Test (units) Treatment Planned Relative Time n H L

Treatment 1 (N=xx)

Source: Listing 16.2.xx

H = Above reference interval, L = Below reference interval

Programming notes: Continued with all tests, treatment groups and time points. The summary is based on the reference ranges (most common ranges used)

Template T\_LB3

Table 14.3.4.xx Summary of laboratory values outside the reference range by treatment

| Laboratory Test (units) | Treatment | m | Н | L | Overall* |
|-------------------------|--------------------|---|---|---|----------|
| | Treatment 1 (N=xx) | | | | _ |

Source: Listing 16.2.xx

H = Above reference interval, L = Below reference interval Subjects only counted once per treatment per category

\*Subjects only counted once per treatment

*m* = total number of results for that parameter

Programming notes: Continued with all tests, treatment groups and time points. The summary is based on the reference ranges (most common ranges used)

13 June 2023 

#### Template T\_LB2

Table 14.3.5.xx Summary of chemistry laboratory values

| | | _ | | • | | • | • | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Test | | Planned | | | | | | | | | | | | |
| (units) | Treatment | Relative Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| | Treatment 1 (N=xx) | | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatments and time points

#### Template T\_UR1

Table 14.3.5.xx Summary of urinalysis results

| | Planned Relativ | e | Treatment : | 1 (N=xx) | Treatment 2 (N=xx) | |
|---|---|---|---|---|---|---|
| Laboratory Test | Time | Result | n | (%) | n | (%) |
| | Time 1 | Positive | Х | х | | |
| | | Negative | X | Χ | | |
| | | Not Done | x | | | |
| | Time 2 | Positive | | | | |
| | | Negative | | | | |
| | | Not Done | | | | |

Source: Listing 16.2.xx

Programming notes: Results recorded as received, e.g. Negative, Trace, etc; urine pH summarised as <5, 5-8, >8; specific gravity summarised as <=1.005, 1.006 - 1.010, 1.011 - 1.015, 1.016 - 1.020, 1.021 - 1.025, 1.026 - 1.029, >=1.030 Continued with all treatment groups and time points. The n's sum to N but the calculated percentages exclude Not Done.

13 June 2023 

#### Template T\_VS1

Table 14.3.6.xx Summary of vital signs

| | | | | | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Planned | | | | | | | | | | | |
| Variable (units) | Treatment | Relative Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median Min | Max |
| Systolic Blood | Treatment 1 (N=xx) | | | | | | | | | | | | |
| Pressure (mmHg) | _ | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all variables, treatments and time points

Column "Variable" isn't required for summary of PBMC data

For PBMC table, add footnote "Note: Results at baseline (Day 1 Pre-dose) are set to 100%"

#### Template T\_VS2

Table 14.3.6.xx Summary of vital signs outside the normal range by treatment, planned relative time and parameter

| | Planned Relative | Systolic Blood<br>Pressure (mmHg) | | Diastolic Blood Pressure (mmHg) | | Heart Rate<br>(beats/min) | | Temperature (C) | | etc | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Time | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Treatment 1 | Time 1 | | | | | | | | | | |
| (N=xx) | Time 2 | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatments and parameters. n = total number of results for that parameter
#### Template T\_VS3

Table 14.3.6.xx Summary of Summary of vital signs outside the normal range by treatment and parameter (excluding baseline time point)

| | Systolic<br>Pressure | | | ic Blood<br>e (mmHg) | | t Rate<br>s/min) | Temper | ature (C) | e | etc | Ove | erall* |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| reatment 1 | | | | | | | | | | | | |

Source: Listing 16.2.xx

Subjects only counted once per treatment per parameter

Programming notes: Continued with all treatments and parameters. n = total number of resul ts for that parameter. Only include post-treatment time points

#### Template T\_EG2

Table 14.3.7.xx Summary of ECG values

| | | | | | | | | | | Cl | nange | from Baseli | ne | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Planned Relative | | | | | | | | | | | | |
| Variable (units) | Treatment | Time | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Heart Rate (bpm) | Treatment 1 (N=xx) | | | | | | | | | | | | | |
| | Treatment 2 (N=xx) | | | | | | | | | | | | | |
| PR Interval (msec) | Treatment 1 (N=xx) | | | | | | | | | | | | | |
| | Treatment 2 (N=xx) | _ | | | | | | | | | | | | |

Source: Listing 16.2.xx

Programming notes: Continued with all treatment groups and time points. Do not summarise RR or QRS axis

13 June 2023 

<sup>\*</sup>Subjects only counted once per treatment

Template T\_EG3

Table 14.3.7.xx Summary of QTcF and PR interval values outside the normal range by treatment, planned relative time and category

| | | | | | ( | QTcF ( | msec) | _ | | | | | PR int. | (msec | <u>) </u> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Planned | | | | | | | >30 | 0-60 | > | 60 | | | | |
| | Relative | 451 | . – 480 | 481 | L – 500 | > | 500 | Incr | ease | Incr | ease | <1 | .20 | >2 | 220 |
| Treatment | Time | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |
| Treatment 1 | Time 1 | | | | | | | | | | | | | | |
| (N=xx) | Time 2 | | | | | | | | | | | | | | |

Source: Listing 16.2.xx

*Programming notes:* Continued with all treatments and time points. n = total number of results for that parameter

Template T\_EG4

Table 14.3.7.xx Summary of QTcF and PR interval values outside the normal range by treatment and category (excluding baseline time point)

| | | | | | Q | TcF (ms | ec) | | | | | PR in | t. (mse | <u>c)</u> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 451 - | - 480 | 481 | - 500 | > | 500 | >30-60 | Increase | >60 | Increase | < | 120 | >2 | 220 | Ove | rall* |
| Treatment | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) | n | (%) |

Source: Listing 16.2.xx

Subjects only counted once per treatment per category

Programming notes: Continued with all treatments and time points. n = total number of results for that parameter. Only include post-treatment time points

13 June 2023 

<sup>\*</sup>Subjects only counted once per treatment

# 19.2.2 Figure Outlines

#### Template F\_PK1

Figure 14.2.xx Individual ASN51 plasma concentration-time plots (linear and semi-log)

Treatment x Day x





Programming notes:

Page by treatment and include all subjects on same page. First page will be Treatment 1 Day 1 followed by Treatment 1 Day 14 before treatment 2

13 June 2023 

#### Template F\_PK2

Figure 14.2.xx Mean (+/- SD) ASN51 plasma concentration-time plots (linear and semi-log)

Day x



Source: Listing 16.2.xx

BQL values are imputed to zero

Programming notes: Page by Day and offset treatment groups (to both sides of timepoint) to minimise overlapping error bars

Remove error bars when producing plots without error bars

13 June 2023 

#### Template F\_PK5

Figure 14.2.xx

Individual ASN51 plasma pre-dose concentration versus day





Source: Listing 16.2.xx

Template F\_PK6

Figure 14.2.xx

Mean (+/- SD) ASN51 plasma pre-dose concentration versus day



Programming notes:

Source: Listing 16.2.xx

Offset treatment groups (to both sides of timepoint) to minimise overlapping error bars

13 June 2023 

#### Template F\_PK10

Listing 16.2.xx Individual ASN51 plasma concentration-time plots for estimation of lambda-z, with regression line



Source: Listing 16.2.xx

13 June 2023 

#### Template F\_SAF1

Figure 14.3.1 Individual systolic blood pressure-time plots

Treatment = Treatment 1 Days 1-13

Programming note: Plots are by treatment groups and Days. Add subject legend. The x-axis label will be "Planned Time Point".

The first page will be "Treatment 1 Days -13" followed by Treatment 1 Day 14 and Follow-up".

Continue with all parameters

13 June 2023 

## **19.2.3** Listing Outlines

Template L\_SD1\_PG

Listing 16.2.x.xx Listing of study dates

Treatment Subject Screening Screening (MRI) Imaging Session 1 Day 1 Day 14 Imaging Session 3 Follow Up

Template L\_SD2\_PG

Listing 16.2.x.xx Listing of reasons for withdrawal

Treatment Subject Date of Withdrawal Study Day Reason

Programming notes: Reason for withdrawal is concatenation of reason and details

Template L\_SD3\_PG

Listing 16.2.x.xx Listing of subjects screened but not enrolled

Screen Number Date of Screen Failure Category Details

Template L\_DV1\_PG

Listing 16.2.x.xx Listing of subjects with inclusion/exclusion criteria deviations

Treatment Subject Type Criterion

Inclusion
Exclusion

13 June 2023 

Template L\_TD1\_PG

Listing 16.2.x.xx Listing of subjects with time deviations

| | | Planned | | | | Time outside the |
|---|---|---|---|---|---|---|
| | | Relative | | Allowed deviation | Actual deviation | deviation window |
| Treatment | Subject | Time | Procedure | (h:min) | (h:min) | (h:min) |

Programming notes: Only include time deviations which exceed the allowed deviation

Template L\_DV2\_PG

Listing 16.2.x.xx Listing of subjects with other protocol deviations

<u>Treatment</u> <u>Subject</u> <u>Protocol Deviation</u> <u>Type of Deviation</u> <u>Category</u>

Template L\_AN1\_PG

Listing 16.2.x.xx Listing of analysis populations

Safety

<u>Treatment</u> <u>Subject</u> <u>Population</u> <u>Population 1</u> <u>Population 2</u> <u>Etc.</u>

13 June 2023 

Template L\_DM1\_PG

Listing 16.2.x.xx Listing of demographic characteristics

| | | | | | | | | | | | Smoking | Cigarettes | Alcohol |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Date of visit | Year of birth | Age (y) | Sex | Race | Ethnicity | Height (cm) | Weight (kg) | BMI (kg/m2) | History | (units) | (units) |
| | | | • | | | | | • | | | | • | |

Treatment 1

Programming notes: A by-subject listing of demographic characteristics including:

Template L\_CM1\_PG

Listing 16.2.x.xx Listing of concomitant medications

| | | | | | | Study Day | | |
|---|---|---|---|---|---|---|---|---|
| | | | | | | Started/ | | |
| | | Medication Class/ | Drug Name/ | Dose/ | Date/time Started/ | Time Since Last | Started Pre- | Ongoing |
| Treatment | Subject | Medication Code* | Indication | Freg/Route | Date Stopped | Dose | Dose? | Medication? |

<sup>\*</sup>Coded using WHOCC ATC/DDD Index vXX.X

Programming notes: Include dose and units (e.g. //Freq/Route

Template L\_MH1\_X

Listing 16.2.x.xx Listing of medical history

| | | | System organ | | Clinical | Date | Date | End relative |
|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Category | class*/Preferred term | Verbatim text | significance | Started | Stopped | to Screening |

<sup>\*</sup>Coded using MedDRA version xx

13 June 2023 

#### Template L\_EX1\_PG

Listing 16.2.x.xx Listing of exposure data

| | | Start Date/ | Stop Date/ | Duration | | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Start Time of Dose | Stop Time of Dose | (days) | Dose | Dose Unit | Formulation/Route | Frequency |
| Treatment 1 | | | | | | | | Once |

Note: Subjects received ASN51 in the fed state on Day 11 only

#### Template L\_PK1\_PG

Listing 16.2.6.xx Listing of ASN51 plasma pharmacokinetic concentration-time data

| | | {Add. | | | | | | <b>Actual Relative</b> | |
|---|---|---|---|---|---|---|---|---|---|
| | | time | | | Planned | Actual time | Time Deviation | Time | |
| Treatment | Subject | var.} | Date | Study Day | Relative Time | (hh:mm) | (min) | (h) | Concentration (units) |

Below the Limit of Quantification (BLQ) is < xx units (e.g. 1 ng/mL)

Programming notes: Values below LLOQ are shown as BLQ. Check LLOQ value in final PK spreadsheet.

#### Template L\_PK4\_PG

Listing 16.2.xx Listing of derived ASN51 plasma pharmacokinetic parameters

| | | | AUC <sub>inf</sub> | $AUC_t$ | $C_{max}$ | t <sub>1/2</sub> | $t_{max}$ |
|---|---|---|---|---|---|---|---|
| Treatment | Subject | Study Day | (units) | (units) | (units) | (units) | (units) |

Programming notes: Continue with all parameters

For Ctrough, report Days across and also include 1 dosing interval after the final dose

13 June 2023 

#### Template L\_PBMC\_PG

Listing 16.2.6.xx Listing of plasma PBMC data

| | | | | Planned | |
|---|---|---|---|---|---|
| Treatment | Subject | Date | Study Day | Relative Time | PBMC pellet (% above baseline) |

Note: Results at baseline (Day 1 Pre-dose) are set to 100%

#### Template L\_AE1\_PG

Listing 16.2.x.xx Listing of all adverse events

| | | | Outcome/ | | | Frequency/ | Related to Study |
|---|---|---|---|---|---|---|---|
| | | System Organ Class*/ | Onset Date/Time/ | Study Day Started/ | Severity/ | Action Taken (1)/ | Drug/ |
| | | Preferred Term/ | Resolved Date/Time/ | Time Since Last | Serious/ | Other Action | Treatment |
| Treatment | Subject | Verbatim Text | Duration | Dose | Withdrawal | Taken | Emergent? |
| Treatment 1 | | Gastrointestinal Disorders / | Resolved/ | Day x/ | Mild/ | Intermittent/ Dose | Possibly/ |
| | | Intestinal Spasm / | | 10d 7h 3m | No/ | not changed/ | Yes |
| | | Intestinal Spasm /<br>Entero-spasm | | 10d 7h 3m | No/<br>Yes | not changed/<br>None | Yes |

(1) Action Taken with Study Treatment \*Coded using MedDRA vXX.X

Programming notes: For the listing of "other significant AEs" include (from ICH E3) AEs leading to withdrawal, AEs leading to dose reduction (including drug withdrawn, interrupted, reduced or similar) and AEs with AEOSE=Y. If AEOSE has not been collected then use "Otherwise significant" in the CRF.

13 June 2023 

#### Template L\_LB1\_PG

Listing 16.2.x.xx Listing of clinical chemistry data outside the normal ranges

| | | | Planned<br>Relative | | Study | | Normal | | Clinically | Reference | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Laboratory test (units) | Time | Date/Time | Day | Value | Interval* | RI | Significant? | Interval# | RI |
| Treatment 1 | | Sodium (mmol/L) | Time 1 | | -1 | 135 | 137 - 145 | L | N | 134 - 142 | |
| | | | Time 2 | | 85 | 143 | 137 - 145 | | | 134 - 142 | Н |
| | | ALT (U/L) | Time 1 | | -1 | 29.00 | 10.0 - 40.0 | | | 10.0 - 40.0 | |
| | | | Time 2 | | 85 | 70.00 | 10.0- 40.0 | Н | Υ | 10.0- 40.0 | Н |

RI for Reference Interval flag, H = Above reference interval, L = Below reference interval

Programming notes: Lists only subjects with at least a high or low value in either of the ranges

#### Template L\_VS1\_PG

Listing 16.2.x.xx Listing of vital signs outside the normal range

| | | | | Systolic | Diastolic | |
|---|---|---|---|---|---|---|
| | | Planned Relative | | <b>Blood Pressure</b> | Blood Pressure | Etc |
| Treatment | Subject | Time | Date/Time | (mmHg) | (mmHg) | (units) |
| | | 24 H | | 63 | 148* | |

<sup>\*</sup> Value outside the normal range

#### Template L\_VS2\_PG

Listing 16.2.x.xx Listing of clinically significant vital signs

| Treatment | Subject | Planned Relative Time | Date/Time | Vital Sign Finding | Comment on Clinical Significance |
|---|---|---|---|---|---|
| <br>- | | | | | |

CS=Clinical Significance

Programming notes: Lists only values with abnormal CS

13 June 2023 

<sup>\*</sup> Used for clinical significance assessment, #Based on most common reference ranges

#### Template L\_EG1\_PG

Listing 16.2.x.xx Listing of QTcF and PR interval values outside the normal range

| QTcF ( | msec) |
|--------|-------|
|--------|-------|

| Planned | | | | Heart Rate | PR Int. | QRS Dur. | QT Int. | | Change from |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | Subject | Relative Time | Date/Time | (bpm) | (msec) | (msec) | (msec) | Observed | Baseline |
| | | 24 H | | 63 | 109* | 78 | 390 | 452* | -6.5 |

#### Template L\_EG2\_PG

Listing 16.2.x.xx Listing of abnormal ECG findings

| Planned Relative | | | | | Comment on Clinical |
|---|---|---|---|---|---|
| Treatment | Subject | Time | Date/Time | ECG Finding | Significance |

*Programming notes:* 

Lists only values with Normal variant='No' or with comment on ECG result

ECG Finding contains Physician's Opinion from CRF and relates to whole trace (not individual parameters), e.g. Normal, Abnormal - NCS or Abnormal - CS

#### Template L\_PE1\_PG

Listing 16.2.x.xx Listing of abnormal physical examination findings

Treatment Subject Planned Relative Time Date Findings Site Details

Treatment 1 Abnormal - NCS

**Programming Notes:** 

List only findings with an 'abnormal' result. Findings is concatenation of result and clinical significance If subjects have multiple abnormal sites at a given time, create a separate row for each site.

13 June 2023 

<sup>\*</sup> Value outside the normal range

#### Template L\_NEURO\_PG

Listing 16.2.x.xx Listing of abnormal neurological examination findings

Treatment Subject Planned Relative Time Date Examination Assessment Findings Details
Treatment 1 Abnormal - NCS

**Programming Notes:** 

List only findings with an 'abnormal' result. Findings is concatenation of result and clinical significance

If subjects have multiple abnormal sites at a given time, create a separate row for each site.

Template L\_CSS\_PG

Listing 16.2.x.xx Listing of positive Columbia-Suicide Severity Rating Scale data

Planned Relative

Treatment Subject Time Date/Time Category Question Result

13 June 2023 

# Appendix A: Laboratory tests with different ranges

| Test | Unit | Sex | Normal ranges* | Reference ranges# |
|---|---|---|---|---|
| Haematocrit | L/L | F | 0.333 – 0.45 | 0.311 – 0.446 |
| Haemoglobin | g/L | F | 113 – 150 | 100 – 150 |
| Lymphocytes | 10^9/L | Both | 1 – 3.4 | 0.9 – 2.84 |
| Mean corpuscular haemoglobin | Pg | Both | 26.1 – 32.7 | 25 – 32.9 |
| Mean corpuscular haemoglobin concentration | g/L | Both | 321 – 355 | 317 – 350 |
| Platelets | 10^9/L | Both | 120 – 326 | 145 – 350 |
| Prothrombin time | sec | Both | 9.4 – 13.5 | 10.2 – 13.9 |
| Sodium | mmol/L | Both | 137 – 145 | 134 – 142 |

<sup>\*</sup> Used for clinical significance assessment, #Based on most common reference ranges

## **Appendix B: Pharmacokinetic analysis**

#### 1 Calculation Methods

## 1.1 Data Handling Conventions

#### 1.1.1 Actual v Planned Times

Actual sample times will be used for the calculation of pharmacokinetic parameters and for individual concentration-time plots.

Planned sampling times will be used to calculate the concentration-time summary statistics and summary concentration-time plots.

#### 1.1.2 Missing and BQL Concentrations

No missing values will be imputed.

For calculation of all pharmacokinetic parameters and individual profile plots, plasma concentrations below the limit of quantification of the assay (BQL) will be treated as missing (except BQL values observed before the maximum concentration, which will be taken as zero).

BQL values will be taken as zero for calculation of plasma concentration summary statistics unless they fall between two quantifiable concentrations in which case they will be treated as missing.

#### 1.2 AUC Calculations

The AUC will be calculated by a combination of linear and logarithmic methods. The linear trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations.

It is acceptable to include data from profiles with >20% extrapolated as long as at least 80% of the profiles in the study have <20% of the  $AUC_{(0-\infty)}$  as extrapolated area. In this instance, individual plasma concentration-time profiles for which the extrapolated areas are >20% of  $AUC_{(0-\infty)}$  will be identified.

It is <u>unacceptable</u> to use  $AUC_{(0-\infty)}$  data if >40% of the AUC has been extrapolated, except in specific situations which should be carefully justified in the study report.

#### 1.3 Lambda-z Calculations

The apparent terminal phase rate-constant ( $\lambda_z$ ) will be estimated by linear regression of logarithmically transformed concentration versus time data. Only those data points which are judged to describe the terminal log-linear decline will be used in the regression.

During the analysis, repeated regressions are carried out using the last three points with non-zero concentrations, then the last four points, last five, etc. Points prior to  $C_{max}$  are not used. Points with a value of zero for the concentration are excluded. For each regression, an adjusted  $R^2$  is computed. The  $\lambda_z$  using the regression with the largest adjusted  $R^2$  is selected. If the adjusted  $R^2$  does not improve, but is within 0.0001 of the largest adjusted  $R^2$  value, the regression with the larger number of points is used.  $\lambda_z$  must be positive, and calculated from at least three data points.

A minimum number of three data points will be used in calculating  $\lambda_z$ .

### 1.4 Observed v Predicted Values

For parameters dependent on  $\lambda_z$ , the 'predicted' rather than the 'observed' parameters will be calculated.

The 'predicted' parameters are calculated using  $\hat{C}_t$  (the predicted value of the concentration at time tn); whilst the 'observed' parameters use the last observed concentration.

# 1.5 Achievement of Steady-State

Achievement of steady state will be judged on the basis of visual interpretation of concentration-time plots.

# 2 Parameter Definitions

# 2.1 Plasma Parameters

| To 4 Combal | D.C.W. | | To dealth do | Log | NN/N/H | CDISC<br>Controlled | TFL |
|---|---|---|---|---|---|---|---|
| Text Symbol | Definition | Calculation | Typical Units | Transform | WNL | Terminology | Symbol |
| | ing and after multiple dosing | T 1 1 4 4 1 1 | /T | V I | | CTROUGH | C . |
| Ctrough | Trough plasma | Trough plasma concentration (measured | ng/mL | Y | - | CIROUGH | $C_{trough}$ |
| | concentration | concentration at the end of a dosing interval | | | | | |
| | | at steady state [taken | | | | | |
| | | directly before next administration, and at 1 | | | | | |
| | | dosing interval after the final dose]) obtained | | | | | |
| | | directly from the concentration-time data. | | | | | |
| | times (Day 1 and after final dos | , , | | | | | |
| C <sub>max</sub> | Maximum (peak) plasma | Obtained directly from the concentration-time | ng/mL | Y | Cmax | CMAX | $C_{max}$ |
| | concentration | data. | | | | | |
| C <sub>max</sub> /Dose | Dose-normalised C <sub>max</sub> | Calculated as C <sub>max</sub> /Dose administered | (ng/mL)/mg | Y | Cmax_D | CMAXD | $C_{max}/D$ |
| t <sub>max</sub> | Time to reach maximum | Obtained directly from the concentration-time | h | N | Tmax | TMAX | t <sub>max</sub> |
| | (peak) plasma concentration | data. | | | | | |
| Half-life (after final | l dose) | | | | | | |
| $\lambda_z$ | Terminal rate constant | Estimated by linear regression of | 1/h | Y | Lambda z | LAMZ | $\lambda_z$ |
| | | logarithmically transformed concentration | | | _ | | |
| | | versus time data. | | | | | |
| t <sub>1/2</sub> | Terminal half-life | Calculated from the terminal slope of the log | h | Y | HL Lambda z | LAMZHL | t <sub>1/2</sub> |
| | | concentration-time curve, as follows: | | | | | |
| | | $\log_e 2$ | | | | | |
| | | $t_{\frac{1}{2}} = \frac{1}{1}$ | | | | | |

13 June 2023 

| Text Symbol | Definition | Calculation | Typical Units | Log<br>Transform | WNL | CDISC<br>Controlled<br>Terminology | TFL<br>Symbol |
|---|---|---|---|---|---|---|---|
| | rve (Day 1 and after final dose) | | | | | | |
| $\mathrm{AUC}_{	au}$ | Area under the plasma concentration-time curve during a dosing interval (t) | Calculated using the trapezoidal method. | h*ng/mL | Y | User specified area | AUCTAU | AUCtau |
| Areas under the cur | rve (after final dose) | | | _ | | | |
| AUC <sub>last</sub> | Area under the plasma<br>concentration-time curve<br>from time zero to time of<br>last measurable<br>concentration | Calculated using the trapezoidal method. | h*ng/mL | Y | AUClast | AUCLST | AUC <sub>last</sub> |
| AUC∞ | Area under the plasma concentration-time curve from time zero to infinity | Calculated using the trapezoidal method for the interval 0 to $t_{last}$ (time $t_{last}$ is the time at which the last non-zero level was recorded), plus the area under the exponential curve from $t_{last}$ to infinity, calculated as follows: $AUC = $ | h*ng/mL | Y | AUCINF_pred | AUCIFP | AUCinf |
| AUC∞/Dose | Dose-normalised AUC∞ | Calculated as AUC <sub>∞</sub> /Dose administered | (h*ng/mL)/mg | Y | AUCINF_D_pred | AUCIFPD | AUC <sub>inf</sub> /D |
| %AUCextrap | Percentage of $AUC_{\infty}$ extrapolated from from $t_{last}$ to infinity | $\%AUC_{extrap} = \frac{100 \times AUC_{t-\infty}}{AUC_{\infty}}$ | % | N | AUC_%EXTRAP_pr<br>ed | AUCPEP | %AUCextrap |
| Clearance and volu | me of distribution (after final do | ose) | | | | | |
| CLss/F | Apparent total clearance from plasma after oral administration | Calculated using the following formula: $CL_{SS} / F = \frac{Dose}{AUC_{\tau}}$ | L/h | Y | Clss_pred (actually derives Clss_F_pred for oral dose) | CLFTAU | CLss/F |
| V <sub>z</sub> /F | apparent volume of<br>distribution after non-<br>intravenous administration<br>calculated at steady state <sup>(3)</sup> | Calculated at steady state will be calculated using the following formula: $V_z/F = \frac{Dose}{\lambda_z \bullet AUC_\tau}$ | L | Y | Vz_pred (actually derives Vz_F_pred for oral dose) | VZFTAU | V <sub>z</sub> /F |
| Accumulation ratio | | | | | | | |
| $R_{ac(AUC)}$ | Accumulation ratio for AUC | Calculated from AUC <sub>t</sub> at steady state and AUC <sub>t</sub> after single dose | - | N | - | ARAUC | R <sub>ac(AUC)</sub> |
| $R_{ac(Cmax)} \\$ | Accumulation ratio for C <sub>max</sub> | $ \begin{array}{c} \text{Calculated from $C_{max}$ at steady state and $C_{max}$} \\ \text{after single dose} \end{array} $ | - | N | - | ARCMAX | Rac(Cmax) |

# Appendix C: Sample page layout

| Asceneuron S.A.: ASN51-103 | | Page x of y |
|---|---|---|
| Population: [Pop] | | |
| | Table [number] [title] | |
| | Column headers | - |
| | Main body of output | - |
| | Source: Listing [16.2.xx] | - |
| Footnotes about the table or listing | ng text go here. | |
| Program: [Prog Name] Produced By: [Username] | [Date] | HMR 22-012 |

Font size will be Arial 9.5pt. The following margins will be used: Left: 1", Right: 1", Top: 1", Bottom: 1"

13 June 2023 

<sup>\*</sup>y = last page of individual output

# ASN51-103 (HMR 22-012) SAP v1.1 (13JUN2023)

Final Audit Report 2023-06-14

Created: 2023-06-13

By:

Status: Signed

Transaction ID: CBJCHBCAABAAahjV94Y7TQdg777F\_ZBRu8J3JkmECYaH

# "ASN51-103 (HMR 22-012) SAP v1.1 (13JUN2023)" History

Document created by

2023-06-13 - 9:32:56 AM GMT- IP address: 31.94.4.197

Document emailed to for signature 2023-06-13 - 9:34:38 AM GMT

1 Email viewed by

2023-06-13 - 9:43:53 AM GMT- IP address: 104.28.124.105

Signer entered name at signing as

2023-06-13 - 4:17:26 PM GMT- IP address: 98.37.192.193

Document e-signed by

Signature Date: 2023-06-13 - 4:17:28 PM GMT - Time Source: server- IP address: 98.37.192.193

Document emailed to for signature

2023-06-13 - 4:17:31 PM GMT

Email viewed by

2023-06-14 - 7:23:29 AM GMT- IP address: 90.243.243.244

Document e-signed by
Signature Date: 2023-06-14 - 7:23:43 AM GMT - Time Source: server- IP address: 90.243.243.244

\_\_\_\_

Document emailed to for signature

2023-06-14 - 7:23:45 AM GMT

🖰 Email viewed by

2023-06-14 - 8:40:10 AM GMT- IP address: 167.98.110.171



Document e-signed by

Signature Date: 2023-06-14 - 8:40:18 AM GMT - Time Source: server- IP address: 167.98.110.171

Agreement completed.

2023-06-14 - 8:40:18 AM GMT